CLINICAL TRIAL: NCT06538623
Title: Single-arm, Open-label Clinical Study of Oxaliplatin Combined With Irinotecan Liposome Injection II Through Hepatic Artery Infusion (HAIC) Followed by 5-Fluorouracil/Leucovorin (HAIC) or Tegorgor Oral Combination Therapy for Hepatic Metastasis of Pancreatic Cancer After First-line Therapy Failure With AG Regimen
Brief Title: Oxaliplatin Combined With Irinotecan Liposome Injection II Through Hepatic Artery Infusion (HAIC) Followed by 5-FU/LV (HAIC) or Tegorgor Oral Combination Therapy for Hepatic Metastasis of Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhongmin Wang, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-246
Record Dates: First submitted 2024-07-31; First posted 2024-08-06 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Neoplasms; Neoplasm Metastasis; Hepatic Metastasis of Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Tegodor 73

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liposome Irinotecan Injection II via Hepatic Arterial Infusion Group (Experimental): Liposome Irinotecan: 60 mg/m², Oxaliplatin: 85 mg/m², Fluorouracil: 2400 mg/m² Leucovorin: 400 mg/m², every 3 weeks (Q3W), administered via hepatic arterial infusion (HAIC); S-1: 40 mg per dose, twice daily for seven days, every 3 weeks (Q3W), taken orally.
  Interventions: Drug: Liposome Irinotecan Injection II combined with Oxaliplatin, Fluorouracil, Leucovorin; Drug: Tegodor

INTERVENTIONS:
Drug: Liposome Irinotecan Injection II combined with Oxaliplatin, Fluorouracil, Leucovorin — Liposome Irinotecan: 60 mg/m², Oxaliplatin: 85 mg/m², Fluorouracil: 2400 mg/m², Leucovorin: 400 mg/m², every 3 weeks (Q3W), administered via hepatic arterial infusion (HAIC);
Drug: Tegodor — Tegodor: 40 mg per dose, twice daily for seven days, every 3 weeks (Q3W), taken orally.

SUMMARY:
The study explores the efficacy and safety of oxaliplatin combined with irinotecan liposome injection II via hepatic arterial infusion (HAIC) followed by sequential treatment with 5-FU/LV (HAIC) or oral administration of S-1 in patients with liver metastasis from pancreatic cancer after the failure of first-line treatment with the AG regimen. This research aims to accumulate more clinical evidence and treatment options for second-line therapy in metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above, with no gender restrictions;
* Pathologically confirmed pancreatic cancer (originating from the pancreatic ductal epithelium), with clinical records indicating metastatic pancreatic cancer, with metastasis limited to the liver;
* Clinical records indicating previous failure of standard AG treatment (having received at least one cycle of standardized chemotherapy, with disease progression or intolerance during treatment, or disease progression after the end of treatment);
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
* Adequate organ function, meeting the following criteria:

  a. Hematological tests:
  1. Neutrophils ≥ 1.5 × 10⁹ /L;
  2. White blood cells ≥ 3.0 × 10⁹ /L;
  3. Platelets ≥ 85 × 10⁹ /L;
  4. Hemoglobin ≥ 70 g/L; b. Biochemical tests:

  <!-- -->

  1. Total bilirubin ≤ 2× upper limit of normal (ULN) (for subjects with biliary obstruction, after biliary drainage ≤ 2.5 × ULN);
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) in metastatic subjects ≤ 5 × ULN;
  3. Albumin level ≥ 28 g/L;
  4. Creatinine clearance rate ≥ 60 ml/min; c. Cardiac function tests:

  <!-- -->

  1. Normal electrocardiogram (ECG) or ECG abnormalities deemed clinically insignificant by the investigator;
  2. Left ventricular ejection fraction (LVEF) ≥ lower limit of normal;
* At least 3 weeks post-surgery, radiotherapy, chemotherapy, or other anti-tumor treatments, with general physical condition or related adverse reactions having recovered (toxicity ≤ grade 1) or stabilized;
* Willing to participate and sign the informed consent form;
* Good compliance and agreement to cooperate with survival follow-up.

Exclusion Criteria:

* Metastatic pancreatic cancer with metastasis to organs other than the liver;
* Subjects with ascites requiring clinical intervention (including moderate to large amounts of ascites; subjects with ascites need to be stable for more than 4 weeks after drainage);
* Clinically severe gastrointestinal diseases (including bleeding, infectious inflammation, perforation, obstruction, or diarrhea greater than grade 1);
* NRS pain score ≥ 4 after standardized treatment with analgesics;
* Second primary malignancy within 5 years (except cured carcinoma in situ, basal cell, or squamous cell skin cancer; subjects with other previous tumors can be enrolled if there has been no recurrence within 5 years);
* Uncontrolled cardiovascular or cerebrovascular diseases with clinical symptoms, including but not limited to: ① NYHA class III or higher heart failure; ② unstable angina; ③ myocardial infarction or stroke within 6 months; ④ supraventricular or ventricular arrhythmias requiring treatment or intervention; ⑤ uncontrolled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg despite optimal treatment);
* Known active hepatitis B subjects (HBsAg positive and HBV DNA ≥ 10³ copies or ≥ 1000 U/ml);
* Active infection or unexplained fever > 38.5°C during the screening period or on the day of administration (subjects with fever caused by tumors can be enrolled as judged by the investigator), which, in the investigator's judgment, would affect the subject's participation in this trial or interfere with the evaluation of efficacy;
* Known allergy to any components of irinotecan hydrochloride liposome, other liposomes, oxaliplatin, 5-FU, LV, or S-1;
* Pregnant or breastfeeding women;
* Women of childbearing potential with a positive blood (urine) pregnancy test during the screening period (both male and female subjects should use reliable contraception during the trial and for 3 months after the last dose to prevent pregnancy);
* Subjects with other medical or social issues that, in the investigator's judgment, might affect their ability to sign informed consent, participation in the trial, or interpretation of the trial results;
* Patients with an estimated survival time of ≤ 3 months are not included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
OS | From enrollment to the death from any cause, assessed up to 18 months
  Overall Survival

SECONDARY OUTCOMES:
ORR | From enrollment to tumor response or date of death from any cause, whichever came first, assessed up to 18 months
  Objective Response Rate (according to RECIST 1.1 criteria)
PFS | From enrollment to tumor progression or date of death from any cause, whichever came first, assessed up to 18 months
  Progression Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wainberg ZA, Melisi D, Macarulla T, Pazo Cid R, Chandana SR, De La Fouchardiere C, Dean A, Kiss I, Lee WJ, Goetze TO, Van Cutsem E, Paulson AS, Bekaii-Saab T, Pant S, Hubner RA, Xiao Z, Chen H, Benzaghou F, O'Reilly EM. NALIRIFOX versus nab-paclitaxel and gemcitabine in treatment-naive patients with metastatic pancreatic ductal adenocarcinoma (NAPOLI 3): a randomised, open-label, phase 3 trial. Lancet. 2023 Oct 7;402(10409):1272-1281. doi: 10.1016/S0140-6736(23)01366-1. Epub 2023 Sep 11. PMID 37708904